CLINICAL TRIAL: NCT06891144
Title: Epidemiological Study of a Prospective Cohort of Patients Aged 60 and Over Managed for Acute Myeloid Leukemia (AML) and Receiving Intensive Induction Therapy
Status: Recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: FILObs_LAMSA 2013
Record Dates: First submitted 2025-03-14; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational epidemiological study targets patients aged 60 and over with de novo or secondary acute myeloblastic leukemia suitable for intensive receive intensive induction therapy as defined by the group. The main aim of the study is to determine the epidemiological characteristics of AML patients, both clinically and biologically, and to correlate these to their outcome. The incidence of AML increases with age, exponentially after the age of 50, giving a median age at diagnosis of close to 70 years, with over half of patients half of patients are over 60 at diagnosis. The principle of treatment as in younger patients, is based on trying to achieve complete remission (CR). remission (CR). Observed complete remission rates range from 38 to 70%. Long-term survival of elderly subjects remains limited, at around 10 to 15%, despite the various types of consolidation tried out in recent years.

years. However, intensive chemotherapy remains the preferred option for initial treatment of these hematological diseases when general condition and comorbidities allow. As shown by Swedish registry studies, it is associated with improved life expectancy.

The proportion of patients who can receive intensive initial treatment is not well known in France, probably varies widely from one region to another, and certainly decreases with increasing age. Only the registry studies currently underway will enable us to assess this precisely.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 and over
* Patients with previously untreated de novo or secondary AML
* Patients suitable for standard intensive treatment
* Patients who have read the information document and agreed to the collection of data concerning them (signature of informed consent).

Exclusion Criteria:

* Patients with AML 3
* Patients with severe, uncontrolled infection at the time of inclusion
* Patients with psychiatric or social disorders that will prevent compliance with the protocol
* Patients without health insurance (affiliation to a social security scheme)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 60 and over with de novo or secondary acute myeloblastic leukemia suitable for intensive induction therapy, as defined by the group's recommendations
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-06 (Actual); Primary Completion 2030-01-06 (Estimated); Study Completion 2031-01-06 (Estimated)

PRIMARY OUTCOMES:
describe the initial characteristics of Acute myeloid leukemia (AML) in patients aged 60 years and older | at diagnosis (from first results related to AML until AML diagnosis) 3 months
  Values for leukocytosis, blasts, neutrophils, and platelets (in /mm3)
describe the initial characteristics of Acute myeloid leukemia (AML) in patients aged 60 years and older | at diagnosis (from first results related to AML until AML diagnosis) 3 months
  the cytogenetic pronosis according ELN criteria
Describe first line AML treatment received | 12 months
  type of treatment
characterize the Overall survival (OS) | 5 years
  defined as the time from date of initiation of chemotherapy to date of death due to any cause. Patients still alive or lost to follow up will be censored at the time they were last known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Pigneux, Prof, Study Chair — French Innovative Leukemia Organization
Locations (27):
- France (27):
  - Angers CHU, Angers
  - Annecy CH, Annecy
  - Avignon CH, Avignon
  - Bayonne CH, Bayonne
  - Besançon CHU, Besançon
  - Brest CHU, Brest
  - CHU Estaing, Clermont-Ferrand
  - Colmar CH, Colmar
  - Grenoble CHU, Grenoble
  - Marseille IPC, Marseille
  - METZ-THIONVILLE CHR- Hôpital de Mercy, Metz
  - Montpellier - Chu Saint Eloi, Montpellier
  - Mulhouse Chu, Mulhouse
  - Nantes CHU, Nantes
  - Nimes CHU, Nîmes
  - Orléans CHU, Orléans
  - Paris Cochin, APHP, Paris
  - Perpignan CH, Perpignan
  - Bordeaux CHU, Pessac
  - Poitiers CHU, Poitiers
  - Reims CHU, Reims
  - Rennes CHU, Rennes
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - ICANS - Institut de cancérologie de strasbourg europe, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - Tours CHU, Tours
  - Nancy CHU, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No